CLINICAL TRIAL: NCT03226028
Title: The Effect of Perioperative Music Listening on Anxiety, Analgesia Use and Patient Satisfaction
Brief Title: Perioperative Music Listening on Anxiety, Analgesia Use and Patient Satisfaction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Sng Ban Leong, Senior Consultant/ Head of Department, Women's Anaesthesia, KK Women's and Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT2017
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Music; Pain; Anxiety; Patient Satisfaction; Analgesia
MeSH Terms: conditions — Pain; Anxiety Disorders; Patient Satisfaction; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music (Experimental): The recruiter will give the patient an ipod with earphone, in which the ipod is equipped with saved playlists of different music genres. Patient will choose the desired playlists and listen to the music for about 30 minutes, seated in a quiet environment in pre-operative waiting area before her turn for the scheduled surgery. Hospital Anxiety and Depression Scale (HADS) and EQ-5D-3L questionnaire will be conducted during this period.
  Patient will be sent to the recovery room after the surgery, and will start the music listening again for 30 minutes once she is ready and feel comfortable to start the session. Pain score, HADS and EQ-5D-3L will be collected from the patient, as well as interview on her satisfaction and experience on the music listening.
  Interventions: Procedure: Music listening

INTERVENTIONS:
Procedure: Music listening — Patient is given an ipod with earphone and with saved playlists of different music genres. Music listening session will be given for 30 minutes before and after surgery. Questionnaires will be asked to fill in. All the earphones will be disinfected following the hospital's infection control guideline.

SUMMARY:
The capacity of music to relieve pain has been used in many forms of medicines and has been proven to reduce anxiety, pain and need for analgesia in perioperative setting. However, music listening as an inexpensive and duplicable method has not been studied in the local context. The investigators hereby propose a prospective study to recruit women who undergo surgery to evaluate the effectiveness of music in pain relief and post-operative recovery in KKH; as well as the possibility of implementing music listening in perioperative setting.

The patients will be offered to listen to one out of several pre-determined lists of music of different genres before, and after surgery. Data including pain score, Hospital Anxiety and Depression Scale (HADS) score, EuroQol-Five Dimensions questionnaire-using Three Levels (EQ-5D-3L), vital signs, analgesia usage and patient satisfaction will be collected in the perioperative period. The collected data shall also be assessed if they are affected by the presence of music, duration of music listening, and the genre chosen by the patients.

The investigators believe that this study could help determine the clinical relevance of music for pain relief in local setting, which potentially could reduce patient pain and anxiety caused by surgery. This in turn could allow music listening to be adopted as a non-invasive pain relief intervention in local healthcare settings and further improve patient outcome with lower cost and greater convenience as well as safety.

DETAILED DESCRIPTION:
Some tissue injury is unavoidable during surgery, but pain and anxiety are (nearly as often) also unavoidable in the perioperative period. Acute post-operative pain and anxiety have been managed via pharmacological interventions such as opioid-based analgesia for over a century. However, non-pharmacological interventions - such as music - have also been shown to safe and cost-effective, to improve the overall patient experience, and improve outcomes across a variety of surgical settings. Music has been shown to decrease pain in the perioperative period, to reduce plasma, urine, and salivary cortisol levels, modulate the inflammatory response (natural killer lymphocytes), blood pressure, and heart rate.Additionally, anxiety scores and pain scores (measured using the visual analog scale (VAS)) have shown statistically significant reductions in the perioperative period, when music therapy was available.

From 1 April 2015 to 31 March 2016, there were 31,871 surgeries done in KK Women's and Children's Hospital (KKH). While music therapy in the hospital has been offered as a part of cognitive rehabilitation services or end of life care, there is little investigation found on its effect if used perioperatively in adult patients who undergo surgeries, especially in local setting. Based on the above rationale, the investigators shall therefore investigate the feasibility and practicability of deploying music listening in pain management in KKH, and further determine the nature of the music (duration, genre) by fitting the local context in order to improve the patient outcome in perioperative settings.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants who are American Society of Anesthesiologists (ASA) 1 and 2 (with well-controlled medical problems);
* Undergo day surgery or same-day-admission gynecologic surgery;
* No hearing impairment.

Exclusion Criteria:

* Patients with significant respiratory disease and obstructive sleep apnea;
* Patients who are unable to read and understand the hospital anxiety questionnaire;
* Obstetric patients.

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only females undergoing gynecologic surgery in KKH will be recruited.
Enrollment: 100 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pain score | Baseline and 1 day
  Difference of Pain score before and after surgery

SECONDARY OUTCOMES:
Change in Analgesia usage | Baseline and 1 day
  Analgesia usage before and after surgery
Change in Patient's satisfaction with the use of music listening | Baseline and 1 day
  Patient's satisfaction on music listening before and after surgery
Change in Hospital Anxiety and Depression Scale (HADS) score | Baseline and 1 day
  HADS Anxiety and Depression score before and after surgery
Change in EQ-5D-3L score | Baseline and 1 day
  EQ-5D-3L score before and after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ban Leong Sng, MBBS, MMED, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tan DJA, Polascik BA, Kee HM, Hui Lee AC, Sultana R, Kwan M, Raghunathan K, Belden CM, Sng BL. The Effect of Perioperative Music Listening on Patient Satisfaction, Anxiety, and Depression: A Quasiexperimental Study. Anesthesiol Res Pract. 2020 Feb 7;2020:3761398. doi: 10.1155/2020/3761398. eCollection 2020. PMID 32089677
- See also: The Effect of Perioperative Music Listening on Patient Satisfaction, Anxiety, and Depression: A Quasiexperimental Study — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7029289/